CLINICAL TRIAL: NCT02387528
Title: Efficacy of a Mindfulness-Based Intervention ("Breathworks for Stress") Versus Relaxation in the Symptoms of Burnout in Primary Care Providers: A Mixed-Methods Pragmatic Controlled Study
Brief Title: Efficacy of a Mindfulness-Based Intervention Versus Relaxation in Primary Care Burnout Providers.
Acronym: MINDFULNESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Daniela D. Sopezki, Phd, Federal University of São Paulo
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CEP639061
Record Dates: First submitted 2015-03-06; First posted 2015-03-13 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Burnout Syndrome
Keywords: MIndfulness; Primary Health Care
MeSH Terms: conditions — Burnout, Psychological | interventions — Mindfulness-Based Stress Reduction; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1- Mindfulness Intervention (Experimental): Mindfulness-Based Intervention: The intervention model tested was "Breathworks for Stress".The mindfulness intervention used in the study had a total of eight encounters, lasting 120 minutes, that took place once a week. In order to accommodate employees' schedule. There was a recommendation of daily practice lasting an average of 15 minutes, as well as the suggestion to use the tools in everyday life.
  In each session a theme was presented, with distinct practices and well-defined objectives
  Interventions: Behavioral: 1- Mindfulness Intervention
- 2- Relaxation Intervention (Placebo Comparator): Relaxation-Based Intervention was composed of four meetings, of two hours duration, held every two weeks. The activities involved mutual help conversations about work situations, psychoeducation on stress and various techniques of stress inoculation, such as: diaphragmatic breathing, progressive muscle relaxation, relaxing visualization and stretching. Each session had its own objective to promote the relaxation response effect.
  Interventions: Behavioral: 2- Relaxation Intervention
- 3- Wait List Control Group (Other): The wait list passive control group did not receive any intervention while the study was been enrolling.
  Interventions: Other: 3- Wait List Control Group

INTERVENTIONS:
Behavioral: 1- Mindfulness Intervention — An intervention program integrating elements of Mindfulness Breathworks Institute Mindfulness based approaches for Pain and illness (MBPI), (Burch , 2009) and Mindfulness Based Stress Reduction (MBSR), (Kabat Zinn, 2003), and Mindfulness based Cognitive Therapy (MBCT) shall be used. All programs are highly structured, lasting eight weeks, with a weekly meeting about two hours , and working with four main techniques during these meetings : mindfulness in breathing, body scan, walking meditation and mindfulness yoga. In order to facilitate the home practice of meditation by participants during and after the intervention protocol, all will receive a CD containing guided meditation sessions, covering the above techniques.
  Other Names: Mindfulness Based Stress Reduction
  Arms: 1- Mindfulness Intervention
Behavioral: 2- Relaxation Intervention — Eight meetings where the participants will practice relaxation techniques.
  Other Names: Relaxation
  Arms: 2- Relaxation Intervention
Other: 3- Wait List Control Group — No intervention
  Other Names: Wait List
  Arms: 3- Wait List Control Group

SUMMARY:
The prevalence of the Burnout Syndrome (BS) or symptoms among Primary Health Care (PHC) providers is high and can affect their quality of life and clinical results. Mindfulness-based interventions (MBI) have been tested as promising interventions to manage chronic stress and BS in PHC providers.

The main goal of this study was to compare the efficacy of an eight week MBI (Group 1 or G1) on burnout symptoms in Brazilian PHC providers, compared to a briefer, four-week relaxation-based intervention (Group 2 or G2) and to a waiting list control group (Group 3 or G3). The initial hypothesis was that the MBI is superior to relaxation and to the waiting list group. A non-randomized controlled trial was performed, with mixed-methods evaluation (qualitative and quantitative).

DETAILED DESCRIPTION:
Study Design: a non-randomized pragmatic controlled trial was performed, with mixed-methods investigation.

Population: The target population of the study were PHC professionals from the city of Porto Alegre in the southern region of Brazil.

Sample: PHC professionals from 50 health units. A sample size calculation was performed, considering an effect size of 0.5 (moderate), with a statistical power of 80% and a confidence interval of 95%. Thus, 65 individuals in each group would be necessary, totaling 195 people distributed in the three groups, estimating a drop-out rate of 10%.

Inclusion criteria: 18 years or over, complete primary education at least, be interested in the objectives of this study and have consented to volunteer to participate in one of the three groups of interventions proposed, being a primary health care worker for at least six months and experiencing any kind of stress in relation to work.

Exclusion criteria: Have been practicing mindfulness, meditation, yoga or similar (tai chi chuan, qi gong) in the last six months, presence of diagnosed clinical diseases that would not allow adherence to the study, being in treatment for psychological or psychiatric problems, in the phase of therapeutic adjustment (less than three months of psychological or pharmacological interventions), be on medical leave of absence from work, dependence or abusive use of alcohol or other drugs, except for tobacco.

Recruitment and procedures: The study was publicized among all PHC units using informative pamphlets, and PHC managers were informed personally by the first author (DS) about the goals of the project. The professionals were dismissed during working hours for the meetings that took place in places available and previously scheduled with the heads of health services. All the volunteers were previously submitted to the study´s criteria for participation. Those who were interested underwent a brief evaluation using the Beck´s Depression Inventory (BDI), Self Reported Questionnaire (SRQ-20) (common mental disorders) and Self Reported Questionnaire (SRQ-A) (alcohol use) scales to exclude severe symptoms (suicidal ideation and alcohol abuse). After inclusion, volunteers were able to choose between the three participant groups of the study (mindfulness, relaxation, or waiting list). We did not randomize the professionals in order to make the study more feasible and pragmatic. Specifically, in a pilot study we had observed that the professionals were highly resistant to being randomly allocated to the study groups.

Ethics: This study was conducted according to the Declaration of Helsinki and was submitted to three Research Ethics Committees, respecting all the criteria for the execution of research with human beings.

All participants agreed to participate in the study and signed the Free and Informed Consent prior to any study procedure.

A drop-out was defined as a participant who completed fewer than four sessions.

Measures:

Added to sociodemographic data, the Maslach Burnout Inventory - General Survey) (MBI-GS ) was used to identify symptoms of BS, The Positive and Negative Scale (PANAS) to evaluate affection, Five Facet Mindfulness Questionnaire (FFMQ) to measure mindfulness dimensions; the Experience Scale to measure decentering and rumination (ES), and the Self-Compassion Scale (SCS) to measure compassion.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers over 18 years old who consent to be randomized to one of two groups, and
* have available time to join the research

Exclusion Criteria:

* Practitioners of mindfulness, meditation yoga or similar in last year,
* presence of not controlled greater severity diseases, such as cancer, schizophrenia, epilepsy, or other psychiatric diseases,
* alcohol or other drugs addiction or abuse, except tobacco, and
* being in acute treatment for psychological or psychiatric problems. All volunteers will undergo a brief initial clinical evaluation to assess whether the conditions of mental and physical health permit participation in groups.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
A mindfulness intervention decreases burnout symptoms | up to 2 months
  Measured by MBI-GS.

SECONDARY OUTCOMES:
A mindfulness intervention decreases negative affect and increases positive affect | up to 2 months
  After the intervention, measured by PANAS
A mindfulness intervention improves self compassion | up to 2 months
  measured by SCE after intervention.
A mindfulness intervention Increases mindfulness state. | up to 2 months
  measured by FFMQ
A mindfulness intervention improves decentering and decrease cognitive rumination | up to 2 months
  Measured by ES - Experience scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Sopezki, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Marcelo Marcos Piva Demarzo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No